CLINICAL TRIAL: NCT00953316
Title: A Prospective Examination of Infant Transition From Car Bed to Car Safety Seat
Brief Title: Infant Transition From Car Bed to Car Safety Seat
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Rhein, Principal Investigator, Boston Children's Hospital
Other Study IDs: X08-03-0176
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Car Seat Transition for At-risk Infants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- at-risk infants: Includes all children born at less than 37 weeks gestation and other high risk newborns such as those with a history of breathing problems and/or low tone.
  Interventions: Other: Measure infant's jaw, record all information about car seat testing, and administer questionnaires.

INTERVENTIONS:
Other: Measure infant's jaw, record all information about car seat testing, and administer questionnaires. — Collect information about car seat testing of infants (until he/she transitions to a car seat), measure the infant's jaw during the first visit using a tape measure 18 different ways by Dr. Rhein or a trained research assistant, and complete a parent questionnaire about car bed use, previous testing of the infant in his/her car seat and information about the infant's home environment such as cigarette smoking, number of other children and daycare arrangements for the infant during the infant's first visit to the clinic. This short questionnaire asks information about car bed use, previous testing of your infant in his/her car seat and information about your home environment such as cigarette smoking, number of other children at your home and daycare arrangements for your infant.

SUMMARY:
This research study has been developed to obtain preliminary information about safe timing of the transition of infants from car beds to car seats, and to find out if initial failure of the car seat challenge is associated with small jaw size or increased respiratory illness.

DETAILED DESCRIPTION:
Studies show that car seats can directly reduce injury in motor vehicle accidents. Unfortunately, some premature and term infants have trouble breathing from the semi-upright seating position in car seats. As a result, the American Academy of Pediatrics recommends car seat challenge testing for at-risk infants, including all children born at less than 37 weeks gestation and other high risk newborns such as those with a history of breathing problems and/or low tone. Infants who fail the car seat test are discharged home in car beds. However, guidelines regarding timing of repeat car seat testing or safe transition back to a car seat are currently unavailable.

At present there is no system for continued evaluation of infants sent home in car beds. In addition, it is not known when it is safe to transition infants from their car bed to a car seat. Infants transitioned too early may still have breathing problems and those transitioned too late may be at risk for injury in the event of a crash. Due to these reasons it is important to find out when it is safe to transition infants from the car bed to a car seat

Moreover, it has recently been shown that some infants with apparent life threatening events (ALTE), have a smaller jaw size than their peers that did not have an ALTE. ALTEs can occur when infants are in their car seats. No studies have been found that looked to see if infants with breathing problems in their car seats also have small jaws. Furthermore no studies have looked to see if infants who fail their initial car seat challenge are at greater risk for respiratory illness during their first year of life.

ELIGIBILITY:
Inclusion Criteria:

* All infants who visit Children's Hospital Boston, Center for Healthy Infant Lung Development for follow up car seat testing

Exclusion Criteria:

* None

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: At-risk infants, including all children born at less than 37 weeks gestation and other high risk newborns such as those with a history of breathing problems and/or low tone.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-04; Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hosptital, Boston, Boston, Massachusetts, United States